CLINICAL TRIAL: NCT03861845
Title: Impact of Pillboxes on Medical Adherence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Florida International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB-18-0451
Record Dates: First submitted 2019-02-27; First posted 2019-03-04 (Actual); Results first posted 2020-08-26 (Actual); Last update posted 2020-08-26 (Actual); Status verified 2020-08

CONDITIONS: Chronic Disease; Medication Adherence
Keywords: Assistive Technology
MeSH Terms: conditions — Chronic Disease; Medication Adherence | interventions — Educational Status

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Standard off-the-shelf pillbox (Active Comparator): Participants will engage in reflection on medication routines. Then they will receive a standard off-the-shelf pillbox. Finally, the participants will receive education & training on how to use the pillbox.
  Interventions: Device: Standard off-the-shelf pillbox; Behavioral: Education & Training; Behavioral: Reflection on medication routines
- Custom off-the-shelf (Experimental): Participants will engage in reflection on medication routines. Then they will receive a custom off-the-shelf pillbox. Finally, the participants will receive education & training on how to use the pillbox.
  Interventions: Device: Custom off-the-shelf pillbox; Behavioral: Education & Training; Behavioral: Reflection on medication routines
- Custom designed and manufactured (Experimental): Participants will engage in reflection on medication routines. Then they will receive a custom designed and manufactured pillbox. Finally, the participants will receive education & training on how to use the pillbox.
  Interventions: Device: Custom designed and manufactured pillbox; Behavioral: Education & Training; Behavioral: Reflection on medication routines

INTERVENTIONS:
Device: Standard off-the-shelf pillbox — Then the participant will receive a store bought one-dose per day pillbox.
  Arms: Standard off-the-shelf pillbox
Device: Custom off-the-shelf pillbox — Then the participant will be administered an off-the-shelf pillbox that was purchased specifically for the participant's preferences, routine, medication regimen, and skills/abilities.
  Arms: Custom off-the-shelf
Device: Custom designed and manufactured pillbox — Then the participant will describe any design preferences for the pillbox. The researcher will design and manufacture the pillbox using a 3D printer, publically available 3D printing object repository, and computer aided design software.
  Arms: Custom designed and manufactured
Behavioral: Education & Training — The participant will receive education and training on how to use the pillbox and how to incorporate the pillbox and taking medications into their daily routine.
Behavioral: Reflection on medication routines — The participant will reflect on his or her daily routine, medication regimen, and use of existing pillboxes. The participant will also engage in a hands-on standardized pillbox task.

SUMMARY:
This study uses an experimental design to test the impact of different types of pillboxes on medication adherence. Participants in this study will randomized to receive one of the three pillbox interventions: 1) A standard seven day a week, one-dose per day pillbox with training 2) an off-the-shelf pillbox that was purchased specifically for the individual's needs with training and education, or 3) a customized 3D printed pillbox that was designed and manufactured specifically to the individual's needs with training and education. Participants will have three visits with the research team to collect baseline data, receive the pillbox, and collect follow up data.

Risks to the study include loss of time, boredom, invasion of privacy, and medication errors. The investigators have taken precautions to mitigate these risks. This study will improve understanding of medication adherence and potentially help us better address poor medication adherence which needlessly causes morbidity, mortality, and costs over $300 million in unnecessary healthcare costs each year.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* speak English
* be prescribed to take two or more medications per day, and manage their own medications.

Exclusion Criteria:

* have a significant cognitive impairment
* unwilling to use a novel pillbox
* unable to meet with the research team

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2019-02-10 (Actual); Primary Completion 2019-05-01 (Actual); Study Completion 2019-05-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jaclyn Schwartz, PhD, Principal Investigator — Florida International University
Locations (1):
- Florida International University, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Schwartz J, Ballard DH. Feasibility of Customized Pillboxes to Enhance Medication Adherence: A Randomized Controlled Trial. Arch Phys Med Rehabil. 2022 Dec;103(12):2288-2295. doi: 10.1016/j.apmr.2022.03.018. Epub 2022 Apr 14. PMID 35430239

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Standard Off-the-shelf Pillbox | Custom Off-the-shelf | Custom Designed and Manufactured
Started | 6 | 5 | 4
Completed | 6 | 5 | 4
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participants enrolled in the study were analyzed. All participants completed the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Off-the-shelf Pillbox | Custom Off-the-shelf | Custom Designed and Manufactured | Total
Number analyzed (Participants) | 6 | 5 | 4 | 15
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: All participants enrolled in the study were analyzed. All participants completed the study.
  Years | 38.50 (20.00) | 46.00 (20.54) | 35.50 (19.05) | 40.20 (19.00)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 0 | 3
  Male | 4 | 4 | 4 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 5 | 4 | 15
  Not Hispanic or Latino | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 5 | 5 | 4 | 14
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 0 | 1
Medication Adherence [Mean (Standard Deviation); unit: units on a scale] — Medication adherence will be measured by the Adherence to Refills and Medications Scale (ARMS). The ARMS is a 7-item assessment. Participants indicate the extent of their adherence on a 4-point Likert-like scale. Scores range from 7 - 28, with higher scores indicating worse medication adherence.
  units on a scale | 11.00 (1.90) | 11.20 (4.49) | 11.50 (1.73) | 11.20 (2.78)

OUTCOME MEASURES:

1. Primary Outcome: Medication Adherence at 1 Month
Description: Medication adherence will be measured by the Adherence to Refills and Medications Scale (ARMS). The ARMS is a 7-item assessment. Participants indicate the extent of their adherence on a 4-point Likert-like scale. Scores range from 7 - 28, with higher scores indicating worse medication adherence.
Time Frame: 1 month
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Standard Off-the-shelf Pillbox | Custom Off-the-shelf | Custom Designed and Manufactured
Number analyzed (Participants) | 6 | 5 | 4
score on a scale | 11.83 (2.71) | 10.20 (2.17) | 9.33 (2.08)

2. Primary Outcome: Satisfaction With Pillbox at 1 Month
Description: The Quebec User Evaluation of Satisfaction with Assistive Technology (QUEST 2.0) quantifies a participant's satisfaction with their pillbox on a five-point Likert-like scale across 8 features (dimensions, weight, ease in opening/closing the device, safety and security, durability, ease of use, comfort, and effectiveness). A score of 1 indicates not satisfied at all and a score of 5 indicates being very satisfied. Scores indicate the average score on the Likert-like scale.
Time Frame: 1 month
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Standard Off-the-shelf Pillbox | Custom Off-the-shelf | Custom Designed and Manufactured
Number analyzed (Participants) | 6 | 5 | 4
score on a scale | 4.65 (0.35) | 4.63 (0.43) | 4.72 (0.28)

3. Secondary Outcome: Number of Participants Who Completed the Study
Description: This metric serves to describe the feasibility of the study and indicates the number of individuals that completed all study interactions. All individuals who enrolled into the study and signed an informed consent document are included in this calculation.
Time Frame: 1 month
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Off-the-shelf Pillbox | Custom Off-the-shelf | Custom Designed and Manufactured
Number analyzed (Participants) | 6 | 5 | 4
Participants | 6 | 5 | 4

ADVERSE EVENTS:
Time Frame: 1 month
Arm/Group | Standard Off-the-shelf Pillbox | Custom Off-the-shelf | Custom Designed and Manufactured
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/5 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/5 | 0/4
Other Adverse Events (participants affected / at risk) | 0/6 | 0/5 | 0/4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Informed Consent Form (2018-12-12): https://cdn.clinicaltrials.gov/large-docs/45/NCT03861845/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2019-02-01): https://cdn.clinicaltrials.gov/large-docs/45/NCT03861845/Prot_SAP_001.pdf